CLINICAL TRIAL: NCT04815850
Title: Phenotyping Seroconversion Following Vaccination Against COVID-19 in Patients on Haemodialysis Study
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: Leicester Hospitals Charity (Other); Francis Crick Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 0810
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2022-05

CONDITIONS: End Stage Kidney Disease
Keywords: haemodialysis; COVID-19; seroconversion; chronic kidney disease
MeSH Terms: conditions — Kidney Failure, Chronic; COVID-19; HIV Seropositivity; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients on haemodialysis: Patients receiving haemodialysis
- Healthy controls: Participants with no chronic kidney disease or history of immunosuppression

SUMMARY:
Patients on haemodialysis are at higher risk of getting a severe form of COVID-19 if they become infected. Vaccinations are soon to arrive and offer great hope of controlling the current pandemic. It is likely that patients on haemodialysis will be amongst the first people to be offered vaccination against COVID-19 when they become available. While any vaccines offered to these patients will be safe to receive, the effectiveness of the vaccines at giving immunity to being infected with COVID-19 are not known as they have not been explicitly tested in patients on haemodialysis. This study will involve having 3 blood tests to test for an antibody response following vaccination for COVID-19. The first will be 1 month after the first vaccination dose to look at the initial antibody response and the second and third will be 1 month and 6 months after the second vaccination dose.

DETAILED DESCRIPTION:
Patients with end stage kidney disease (ESKD) on haemodialysis are more likely to suffer poorer outcomes following infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. This is likely to be because these patients have higher levels of co-morbid diseases and they are relatively immunosuppressed due to the effects of advanced kidney disease. The humoral response against common viral vaccination is known to be blunted in patients with ESKD and there are data to suggest seroconversion following infection with COVID-19 is blunted in patients with kidney disease. A successful programme of vaccination will undoubtedly improve outcomes for patients on haemodialysis, but vaccine testing programmes have not included patients with ESKD. Whilst initial press-coverage of the efficacy of vaccines which are available for use is promising, they are untested in patients on haemodialysis who are known to be relatively immunosuppressed as a result of their renal disease and as such the efficacy for this patient group is not known.

This study will phenotype the IgG antibody response to vaccination for COVID-19 in 100 patients on haemodialysis compared to 50 healthy volunteers. Antibody testing will be conducted at 1 month post first vaccination dose and 1 month and 6 months post second vaccination dose. This will give crucial information as to the efficacy of the vaccine and inform possible requirements for re-vaccination.

This study will:

1. Phenotype the 1 month IgG antibody response to the first vaccination dose and the 1 month and 6 month response to the second vaccination dose for COVID-19 in patients on haemodialysis
2. Compare the 1 month IgG antibody response to the first vaccination dose and the 1 month and 6 month response to the second vaccination dose for COVID-19 between patients on haemodialysis and healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* End stage kidney disease on haemodialysis
* Able and willing to give informed consent
* Have completed or due to complete vaccination against COVID-19

Exclusion Criteria:

* Acute kidney injury requiring temporary haemodialysis
* Unable to give informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving haemodialysis at Leicester General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew PM Graham-Brown, Principal Investigator — University of Leicester
Locations (1):
- University Hospital Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients on Haemodialysis
Started | 94
Completed | 94
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients on Haemodialysis
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in COVID-19 IgG Antibody (Relative Light Units)
Description: Measured from a serum blood sample. Serum was tested for the presence of SARS-CoV-2 neutralising IgG and IgM antibodies directed against the receptor binding domain of the S1 spike protein, using the Siemens ADVIA Centaur XP/XPT assay and reported as positive or negative as per manufacturer guidelines (detectable antibody levels >1RLU (relative light units) reported as positive to an upper limit of 10)
Time Frame: 1 month post first vaccine
Measure: Median (Standard Error); unit: relative light unit (RLU)
Arm/Group | Patients on Haemodialysis
Number analyzed (Participants) | 94
relative light unit (RLU) | 2.4 (8.8)

ADVERSE EVENTS:
Time Frame: 10 months
Description: This is an observational study. There were no adverse events related to the study procedures which involved blood samples and questionnaires.
Arm/Group | Patients on Haemodialysis
All-Cause Mortality (participants affected / at risk) | 29/94
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT04815850/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04815850/SAP_001.pdf